CLINICAL TRIAL: NCT07381777
Title: Phase II Randomized Trial of XELOX Plus DoSTARlimab Versus XELOX Alone as Consolidation Treatment After Standard Chemoradiation in pMMR/MSS or MSI-Low Locally Advanced Rectal Cancer (LARC) Patients - IMMUNOSTAR Trial GOIRC-02-2024
Brief Title: XELOX Plus DoSTARlimab Versus XELOX Alone as Consolidation Treatment After Standard Chemoradiation in pMMR/MSS or MSI-Low Locally Advanced Rectal Cancer (LARC) Patients
Acronym: IMMUNOSTAR
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOIRC-02-2024
Record Dates: First submitted 2025-03-28; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-05

CONDITIONS: Locally Advanced Rectal Cancer (LARC)
Keywords: Consolidation chemotherapy; dostarlimab; pMMR/MSS; MSI-Low; LARC; phase II; clinical complete response (cCR); safety
MeSH Terms: interventions — XELOX; Capecitabine; Oxaliplatin; dostarlimab

STUDY DESIGN:
Intervention Model Description: randomization (2:1) to consolidation chemotherapy (XELOX) plus anti-PD-1 antibody (dostarlimab) after standard long-course CRT followed by adjuvant dostarlimab VS follow-up (ARM A) compared to XELOX alone as consolidation (ARM B) Arm A subsequent randomization (1:1) to adjuvant dostarlimab for a maximum of 8 cycles (ARM A1) VS only follow-up (ARM A2), and in ARM B only follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XELOX + DOSTARLIMAB (Arm A) (Experimental): 4 cycle - consolidation chemotherapy (XELOX) plus anti-PD-1 antibody (dostarlimab) after standard long-course CRT, followed by randomisation to adjuvant dostarlimab (Arm A1) versus follow-up (Arm A2)
  Interventions: Drug: XELOX (Capecitabine and Oxaliplatin); Drug: Dostarlimab
- XELOX (Arm B) (Active Comparator): 4 cycle- XELOX alone as consolidation treatment
  Interventions: Drug: XELOX (Capecitabine and Oxaliplatin)

INTERVENTIONS:
Drug: XELOX (Capecitabine and Oxaliplatin) — Capecitabine 1000mg/m2 BID + Oxaliplatin 130mg/m2 Q3W
Drug: Dostarlimab — Dostarlimab IV 500mg Q3W
  Arms: XELOX + DOSTARLIMAB (Arm A)

SUMMARY:
This is a phase II, multicenter, randomized (2:1) controlled, clinical trial to evaluate the preliminary efficacy and safety of consolidation chemotherapy (XELOX) plus dostarlimab after standard long-course CRT (ARM A) compared to XELOX alone (ARM B) in patients with pMMR/MSS or MSI-Low LARC (cT3-4 cN0, any cT cN+) candidate to receive standard long course CRT followed by TME. After the surgery, the patients in ARM A will be randomized (1:1) to receive adjuvant dostarlimab (ARM A1) versus follow-up (ARM A2), and in ARM B only follow-up.

If clinical complete responses (cCR) are documented after consolidation treatment, the patient may choose not to proceed with surgery and pursue nonoperative management (NOM).

DETAILED DESCRIPTION:
This is a phase II, multicenter, randomized (2:1) controlled, clinical trial to evaluate the preliminary efficacy and safety of consolidation chemotherapy (XELOX) plus anti-PD-1 antibody (dostarlimab) after standard long-course CRT followed by adjuvant dostarlimab versus follow-up (ARM A) compared to XELOX alone as consolidation (ARM B) in patients with pMMR/MSS or MSI-Low LARC (cT3-4 cN0, any cT cN+) candidate to receive standard long course CRT followed by TME.

Subsequent randomization into a ratio 1:1 will be performed after surgery, only for patients randomized in ARM A, to receive adjuvant dostarlimab for a maximum of 8 cycles (ARM A1) versus only follow-up (ARM A2), and in ARM B only follow-up (Figure 1).

If clinical complete responses (cCR) are documented after restaging, the patient may choose not to proceed with surgery and pursue nonoperative management (NOM) (Figure 1).

The patients before randomization will be stratified as follows:

* cT4 or < cT4 stage;
* positive or negative lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven rectal adenocarcinoma with distal extension less 16 cm from the anal verge.
* Stage cT3-4 cN0 cM0, any cT cN+ M0 [N+ stage, three or more lymph nodes of diameter >0.5 cm measured by endorectal ultrasound, or one or more lymph nodes of diameter >1 cm measured by magnetic resonance (MRI)].
* Proficient mismatch repair (pMMR)/microsatellite stable status (MSS) or microsatellite instability (MSI)-low (MSI-L)
* ECOG-Performance Status 0-1
* No previous treatment with chemotherapy or radiation therapy.
* No prior exposure to immune-mediated therapy, excluding therapeutic anticancer vaccines.
* Neutrophil count >1,500/mL, platelet count >100.000/mL, hemoglobin >9.0 g/dL, serum creatinine <1.5 3 upper limit of normal (ULN), alanine aminotransferase and aspartate aminotransferase 2.5 3 ULN, total bilirubin <1.5 3 ULN.
* Signed written informed consent.

Exclusion Criteria:

* Subjects with active, known, or suspected autoimmune disease requiring systemic treatment (systemic steroids or immunosuppressive agents), except for subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune conditions only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Distant metastases documented.
* Participants have received a live vaccine within 30 days of the planned start of study therapy. COVID-19 vaccines that do not contain live viruses are allowed. Note: mRNA and adenoviral-based COVID-19 vaccines are considered non-live.
* Participants have a current active history of pneumonitis or interstitial lung disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response (cCR) at 12 months | After 12 months of the end of the consolidation therapy
  To evaluate the clinical complete response (cCR) after 12 months of the end of consolidation treatment, defined as an absence of residual disease on digital and endoscopic rectal examination, as well as the absence of residual disease on rectal MRI, with no restricted diffusion on T2-weighted imaging (cT0N0M0), or the pathological complete response (pCR), in patients who undergo surgery, defined as an absence of viable tumor cells after full pathologic examination of the resected specimen (pT0N0M0)

SECONDARY OUTCOMES:
Clinical complete response (cCR) at 24 and 36 months | After 24 and 36 months of the end of the consolidation therapy
  To evaluate cCR at 24 and 36 months defined as an absence of residual disease on digital and endoscopic rectal examination, as well as the absence of residual disease on rectal MRI, with no restricted diffusion on T2-weighted imaging
Assessment of Organ Preservation Rate | From the enrollmentat to any time up to 3 years
  To assess Organ Preservation Rate defined as not undergoing Total Mesorectal Excision (TME), either as primary management or for local recurrence, or who did not have a permanent colostomy created, at any time up to 3 years.
Disease Free Survival | From randomization to recurrence of a tumor up to 3 years
  To evaluate DFS
Overall Survival | From initiation of study treatment to death from any cause up to 3 years
  To evaluate OS
Pathological Downstaging Rate | Perioperative period (at surgical resection).
  Pathological downstaging defined as a reduction in tumor stage comparing post-surgical pathological TNM stage (ypTNM) with baseline clinical TNM stage (cTNM).
Improvement of Quality of Life | Baseline, during treatment, and at the end of adjuvant therapy (approximately 12 months).
  To assess the QoL measured as pre-defined PRO endpoints in this study are mean changes from baseline in the EORTC-QLQ-CR29 questionnaire administered at baseline, after chemoradiation, after consolidation therapy, before to start adjuvant therapy and at the end of adjuvant therapy
Adverse Events | From first dose of study treatment through study completion, an average of 3 years
  To evaluate safety in terms of incidence, nature, frequency and severity of Adverse Events (AEs) and laboratory abnormalities graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v.5.0.
Association Between ctDNA Status and Clinical Outcomes | From ctDNA assessment during treatment through follow-up, up to 3 years.
  ctDNA status (positive vs negative) assessed at predefined time points and its association with clinical outcomes, including disease recurrence and treatment decisions.

CONTACTS AND LOCATIONS:
Locations (30):
- Italy (30):
  - Ospedale San Donato - UOC Oncologia Medica dell'Aretino, Casentino, Valtiberina, Valdichiana Aretina, Arezzo
  - Oncologia medica e prevenzione oncologica - Centro di Riferimento Oncologico, Aviano
  - UOC Oncologia Medica IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - Oncologia Medica Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - UOC Oncologia Medica - ARNAS Garibaldi PO Nesima, Catania
  - A.O. Oncologia S. Croce e Carle - presidio Ospedaliero A. Carle, Cuneo
  - AOUC Azienda Ospedaliero - Universitaria Careggi Oncologia Medica, Florence
  - U.O. Oncologia Medica 1 IRCCS Ospedale Policlinico San Martino, Genova
  - S.C. Oncologia Medica, Ospedale Felettino, La Spezia
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola (FC)
  - Oncologia Falck - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Struttura Complessa Oncologia Medica 1 - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - AOU di Modena - Policlinico di Modena - DH Oncologico, Modena
  - Oncologia Clinica Sperimentale Addome Istituto Nazionale Tumori - IRCCS Fondazione G. Pascale, Napoli
  - UOC Di Oncologia Medica AOU Federico II, Napoli
  - UOC Oncoematologia AOU Vanvitelli, Napoli
  - UOC Oncologia 1 - Ospedale Busonera - IRCCS Istituto Oncologico Veneto, Padua
  - UOC Oncologia Medica Azienda Ospedaliero Universitaria di Parma, Parma
  - SC Oncologia, Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Oncologia Medica 2 Universitaria, Pisa
  - UOC Oncologia Ravenna Dipartimento di Oncologia ed Ematologia - AUSL Romagna, Ravenna
  - SOC di Oncologia Provinciale, AUSL IRCCS di Reggio Emilia, Reggio Emilia
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma
  - Oncologia Medica - Policlinico Universitario Gemelli IRCCS, Roma
  - IRCCS Istituto clinico humanitas, Rozzano
  - Oncologia Ricerca Clinica - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - U.O. C. di Oncologia Medica - OSPEDALE CIVILE SS ANNUNZIATA, Sassari
  - Oncologia Medica 1, A.O.U. Città della Salute e della Scienza di Torino Ospedale Molinette, Torino
  - SOC Oncologia Azienda sanitaria Universitaria Friuli Centrale - P.O. S. Maria della Misericordia, Udine
  - ASST Brianza, Vimercate